CLINICAL TRIAL: NCT00623350
Title: Stroke Team Remote Evaluation Using a Digital Observation Camera Arizona - The Initial Mayo Clinic Experience
Brief Title: Stroke DOC Arizona TIME - Stroke Team Remote Evaluation Using a Digital Observation Camera
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Arizona Department of Health Services (Other Government); Yuma Regional Medical Center (Other); Kingman Regional Medical Center (Other); University of California, San Diego (Other)
Responsible Party: Bart Demaerschalk, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-005731
Record Dates: First submitted 2008-02-15; First posted 2008-02-26 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Stroke, Acute
Keywords: Telemedicine; Stroke, Acute; Rural; Thrombolysis; Consultation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Acute Stroke Telephone consult for the decision of tPA within 3 hours of symptoms onset.
  Interventions: Other: Telephone
- 2 (Active Comparator): Acute Stroke consult via audio video telemedicine for the decision of tPA within 3 hours of symptom onset.
  Interventions: Other: Two way audio/video telemedicine consult

INTERVENTIONS:
Other: Telephone — Acute Stroke consult by Telephone for the decision of tPA within 3 hours of symptom onset.
  Arms: 1
Other: Two way audio/video telemedicine consult — Acute Stroke consult by two way audio video telemedicine for the decision of tPA within 3 hours of symptom onset.
  Arms: 2

SUMMARY:
Noninvasive prospective multi-center study of an interactive 2-way, wireless or site-independent, audiovisual telemedicine system designed for real-time remote examination of acute stroke symptoms and deficits as a basis for treatment consultation and recommendation.

Study aims (1) to determine the impact of a site-independent, remote, telemedicine consultation system on decision making in the Emergency Department, regarding the decision to treat or not to treat with thrombolytics; (2) to assess the numbers of patients who receive thrombolytics and the time to treatment in patients evaluated by telemedicine versus telephone only; (3) to assess the appropriateness of thrombolytic treatment decisions in telemedicine versus telephone-only consultations; and (4) to assess the completeness of the data collection in telemedicine versus telephone-only consultations.

60 patients in Arizona with acute presentation of stroke symptoms, per bedside practitioner discretion (onset generally less than 12 hours and likely less than 3 hours)

Two arms: Video Camera/Telemedicine (Intervention n = 30) and No Video Camera/Telephone only (Control n = 30)

DETAILED DESCRIPTION:
Design

Noninvasive prospective multi-center study of an interactive 2-way, wireless or site-independent, audiovisual telemedicine system designed for real-time remote examination of acute stroke symptoms and deficits as a basis for treatment consultation and recommendation.

Study aims (1) to determine the impact of a site-independent, remote, telemedicine consultation system on decision making in the Emergency Department, regarding the decision to treat or not to treat with thrombolytics; (2) to assess the numbers of patients who receive thrombolytics and the time to treatment in patients evaluated by telemedicine versus telephone only; (3) to assess the appropriateness of thrombolytic treatment decisions in telemedicine versus telephone-only consultations; and (4) to assess the completeness of the data collection in telemedicine versus telephone-only consultations.

60 patients in Arizona with acute presentation of stroke symptoms, per bedside practitioner discretion (onset generally less than 12 hours and likely less than 3 hours)

Two arms: Video Camera/Telemedicine (Intervention n = 30) and No Video Camera/Telephone only (Control n = 30)

Assessments

All cases will undergo the following assessments:

Patient-Level Visits

Baseline: Pre-stroke Modified Rankin Scale (demographics), pre-treatment Modified Rankin Scale, medications during prior 3 days, physical exam and vital signs, NIHSS, Modified NIHSS, EKG, screening labs, and head CT scan

Treatment: Treatment times, thrombolytic safety outcome, and recanalization treatment

Day 90: Modified Rankin Scale, Barthel Index, and mortality

End of Study: End of study/Termination

Meta-Level Reviews

Adjudication: Post case completion, review and evaluation of each remote consultation on whether the recommendation for or against thrombolytic therapy was appropriate, given the information presented at each of 3 levels of adjudication.

Central Read: Post case completion, review and evaluation of each Baseline head CT scan interpretation on whether there was a CT contraindication to thrombolytic therapy.

Trial Groups

There will be two trial groups in this study. The investigators hypothesized (based upon sample size calculations) that the correct treatment will be recommended at rates of 80% (telephone) and 90% (full telemedicine).

Target Population

60 AZ patients will be randomized to either telephone-only or video telemedicine consultation. Appropriateness of therapeutic decision-making, numbers treated, time to treatment, and completeness of data collection will be evaluated and compared for each group.

If the protocol or grant application is investigator-initiated, a 200-word (or less) abstract of the proposed protocol or grant application must be included (an abstract included in an NIH or other submission is acceptable). If the protocol is sponsor initiated, a summary written by the Mayo investigator must be included. Summary should include: 1) Hypothesis, 2) Basic study plan, 3) Statistical method/rationale, 4) Scientific basis or justification, 5) Inclusion/exclusion criteria, and 6) Monetary consideration. You may type or cut and paste from an existing document to address this question

Objectives

1. to determine the impact of a site-independent, remote, telemedicine consultation system on decision making in the Emergency Department, regarding the decision to treat or not to treat with thrombolytics;
2. to assess the numbers of patients who receive thrombolytics and the time to treatment in patients evaluated by telemedicine versus telephone only;
3. to assess the appropriateness of thrombolytic treatment decisions in telemedicine versus telephone-only consultations; and
4. to assess the completeness of the data collection in telemedicine versus telephone-only consultations.

ELIGIBILITY:
Subject Inclusion Criteria

For inclusion in the study, subjects must fulfill all of the following criteria:

* Written Informed Consent
* Eighteen years of age or older
* Symptoms consistent with acute stroke (ischemic or hemorrhagic)
* Acute presentation of stroke symptoms, per bedside physician discretion (onset generally less than 12 hours and likely less than 3 hours)

Subject Exclusion Criteria

The following is the sole criterion for exclusion from the study:

* Unlikely to complete study through 90-day follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-12; Primary Completion 2008-11 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
to determine the impact of a site-independent, remote, telemedicine consultation system on decision making in the Emergency Department, regarding the decision to treat or not to treat with thrombolytics | 90 days
to assess the numbers of patients who receive thrombolytics and the time to treatment in patients evaluated by telemedicine versus telephone only | 90 days
to assess the appropriateness of thrombolytic treatment decisions in telemedicine versus telephone-only consultations | 90 days
to assess the completeness of the data collection in telemedicine versus telephone-only consultations. | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Phoenix, Arizona, United States

REFERENCES:
- [Result] Demaerschalk BM, Bobrow BJ, Raman R, Kiernan TE, Aguilar MI, Ingall TJ, Dodick DW, Ward MP, Richemont PC, Brazdys K, Koch TC, Miley ML, Hoffman Snyder CR, Corday DA, Meyer BC; STRokE DOC AZ TIME Investigators. Stroke team remote evaluation using a digital observation camera in Arizona: the initial mayo clinic experience trial. Stroke. 2010 Jun;41(6):1251-8. doi: 10.1161/STROKEAHA.109.574509. Epub 2010 Apr 29. PMID 20431081
- [Derived] Demaerschalk BM, Bobrow BJ, Raman R, Ernstrom K, Hoxworth JM, Patel AC, Kiernan TE, Aguilar MI, Ingall TJ, Dodick DW, Meyer BC; Stroke Team Remote Evaluation Using a Digital Observation Camera (STRokE DOC) in Arizona-The Initial Mayo Clinic Experience (AZ TIME) Investigators. CT interpretation in a telestroke network: agreement among a spoke radiologist, hub vascular neurologist, and hub neuroradiologist. Stroke. 2012 Nov;43(11):3095-7. doi: 10.1161/STROKEAHA.112.666255. Epub 2012 Sep 13. PMID 22984007
- [Derived] Demaerschalk BM, Raman R, Ernstrom K, Meyer BC. Efficacy of telemedicine for stroke: pooled analysis of the Stroke Team Remote Evaluation Using a Digital Observation Camera (STRokE DOC) and STRokE DOC Arizona telestroke trials. Telemed J E Health. 2012 Apr;18(3):230-7. doi: 10.1089/tmj.2011.0116. Epub 2012 Mar 8. PMID 22400970
- [Derived] Miley ML, Demaerschalk BM, Olmstead NL, Kiernan TE, Corday DA, Chikani V, Bobrow BJ. The state of emergency stroke resources and care in rural Arizona: a platform for telemedicine. Telemed J E Health. 2009 Sep;15(7):691-9. doi: 10.1089/tmj.2009.0018. PMID 19694588
- [Derived] Capampangan DJ, Wellik KE, Bobrow BJ, Aguilar MI, Ingall TJ, Kiernan TE, Wingerchuk DM, Demaerschalk BM. Telemedicine versus telephone for remote emergency stroke consultations: a critically appraised topic. Neurologist. 2009 May;15(3):163-6. doi: 10.1097/NRL.0b013e3181a4b79c. PMID 19430275
- [Derived] Demaerschalk BM, Miley ML, Kiernan TE, Bobrow BJ, Corday DA, Wellik KE, Aguilar MI, Ingall TJ, Dodick DW, Brazdys K, Koch TC, Ward MP, Richemont PC; STARR Coinvestigators. Stroke telemedicine. Mayo Clin Proc. 2009;84(1):53-64. doi: 10.4065/84.1.53. PMID 19121244